CLINICAL TRIAL: NCT04966299
Title: Effect of Daily Erythritol Versus Sucrose Intake Over 5 Weeks on Glucose Tolerance in Adolescents: a Pilot Trial
Brief Title: Effect of Daily Erythritol Versus Sucrose Intake Over 5 Weeks on Glucose Tolerance in Adolescents
Acronym: EryAdo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EryAdo
Record Dates: First submitted 2021-05-25; First posted 2021-07-19 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Insulin Resistance; Glucose Tolerance; Body Composition; Gastrointestinal Tolerance; Thrombocyte Aggregation; Blood p-Selectin; Blood Erythritol; Blood Xylitol
MeSH Terms: conditions — Insulin Resistance | interventions — Sucrose; Glucose; Fructose; Xylitol; Water

STUDY DESIGN:
Intervention Model Description: EryClot-Pilot:
  This trial is a randomized, double-blind, crossover trial. The project set-up is single-center, national. In total, 3 volunteers will be enrolled. There will be 3 study arms.
  EryClot This trial is a randomized single-blind, crossover trial. The project setup is single-center national. In total 10 volunteers will be enrolled. There will be 3 study arms.
  EryClot in vitro This trial is an in vitro trial using human blood samples. The project setup is single-center national. In total blood samples from 12 volunteers will be collected.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Sucrose (Active Comparator): 15 participants receive 25g sucrose per day during 5 weeks
  Interventions: Dietary Supplement: Sucrose
- Erythritol (Experimental): 15 participants receive 36g eryhtritol per day during 5 weeks
  Interventions: Dietary Supplement: Eryhtritol
- EryClot-Pilot Erythritol (Experimental): 3 participants receive 50g erythritol dissolved in 300mL water once during the visit
  Interventions: Dietary Supplement: Eryhtritol
- EryClot-Pilot Glucose (Active Comparator): 3 participants receive 75g glucose dissolved in 300mL water once during the visit
  Interventions: Dietary Supplement: Glucose
- EryClot-Pilot Fructose (Active Comparator): 3 participants receive 25g fructose dissolved in 300mL water once during the visit
  Interventions: Dietary Supplement: Fructose
- EryClot Erythritol (Experimental): 10 participants receive 50g erythritol dissolved in 300mL water once during the visit
  Interventions: Dietary Supplement: Eryhtritol
- EryClot Xylitol (Experimental): 10 participants receive 33.5g xylitol dissolved in 300mL water once during the visit
  Interventions: Dietary Supplement: Xylitol
- EryClot Water (Placebo Comparator): 10 participants receive 300mL water once during the visit
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Eryhtritol — Eryhtritol-sweetened beverages twice a day (36g erythritol/day) with main meals during 5 weeks
  EryClot-Pilot:
  Erythritol 50g dissolved in 300mL water administered once per visit
  EryClot:
  Erythritol 50g dissolved in 300mL water administered once per visit
  Other Names: E968-Erythritol
  Arms: EryClot Erythritol; EryClot-Pilot Erythritol; Erythritol
Dietary Supplement: Sucrose — Sucrose-sweetened beverages twice a day (25g sucrose/day) with main meals during 5 weeks
  Arms: Sucrose
Dietary Supplement: Glucose — Glucose 75g dissolved in 300mL water administered once per visit
  Arms: EryClot-Pilot Glucose
Dietary Supplement: Fructose — Fructose 25g dissolved in 300mL water administered once per visit
  Arms: EryClot-Pilot Fructose
Dietary Supplement: Xylitol — Xylitol 33.5g dissolved in 300mL water administered once per visit
  Other Names: E967-Xylitol
  Arms: EryClot Xylitol
Dietary Supplement: Water — 300mL water administered once per visit
  Arms: EryClot Water

SUMMARY:
Childhood and adolescence are crucial periods for prevention of obesity, as obese children are five times more likely to be obese at adulthood than lean children. To this purpose, sugar consumption should be reduced. The sugar alcohol erythritol is increasingly popular as sugar substitute in the food industry and is also recommended to diabetic patients. The substance is freely available. Recent acute studies show that erythritol has a positive influence on satiation and gastric emptying without affecting insulin and plasma glucose. In this trial, the investigators aim to assess the effect of a chronic intake of erythritol versus sucrose on insulin resistance in healthy adolescents.

EryClot-Pilot:

Erythritol is also produced by the human body and possibly elevated erythritol levels in the blood are an indication of an increased risk of cardiovascular disease, obesity or diabetes in the future.

In a recently published study, a possible effect of erythritol on blood clotting function was described. In this in vitro experiment, increased blood clotting was observed when erythritol was added to clotting cells (platelets) in the test tube. Studies in humans on blood coagulation after administration of erythritol are missing so far.

With a pilot study, the investigators study whether erythritol is detectable in the blood after administration of glucose and fructose. Furthermore, the erythritol level in the blood and a possible effect on the blood coagulation function after administration of erythritol will be investigated.

These preliminary tests serve to clarify the data situation so that further studies can be based on them.

The preliminary results of the EryClot_Pilot study indicate that there appears to be no measurable effect of erythritol on thrombocyte aggregation. This implicates that there is a discrepancy between our results and the results reported in a recent published study. This is why we need to assess the effects of erythritol administration on more parameters of blood coagulation as well as in more subjects.

Due to a study published in June 2024, there appears the need to investigate the effects of xylitol on blood clotting function as well.

EryClot in vitro:

In addition to the human EryClot study, we will conduct in vitro experiments (aggregometry assay after addition of erythritol or xylitol in human platelet rich plasma).

DETAILED DESCRIPTION:
This trial aims to assess the effects of the daily intake of an erythritol-sweetened beverage over 5 weeks on insulin resistance, glucose tolerance and metabolism as well as on gut microbiota. Moreover, this study will also assess the effect of the above-mentioned intervention on food intake, body composition and gastrointestinal tolerance in this population.

EryClot-Pilot:

The aim of this pilot study is to investigate whether erythritol is detectable in the blood after administration of glucose and fructose. Furthermore, the erythritol level in the blood and a possible effect on the blood clotting function after administration of erythritol will be investigated.

EryClot:

The aim of this study is to investigate the erythritol level in blood after administration of erythritol and a possible effect on blood clotting function. Additionally, a possible effect of xylitol on blood clotting function will be investigated.

EryClot in vitro:

The aim of this study is to investigate the platelet responsiveness in vitro in human plasma after addition of erythritol and xylitol.

ELIGIBILITY:
EryAdo:

Inclusion Criteria:

* Healthy adolescents
* Aged 14-18 years
* Normal weight (BMI between 15th and 85th percentile for age and gender)
* Minimum weight of 45kg
* Regular sugar consumption >25g/d

Exclusion Criteria:

* Severe acute or chronic diseases
* Pregnancy
* Regular intake of prebiotics
* Regular intake of probiotics
* Regular intake of pro-/prebiotic foods
* Antibiotics cure within 3 months preceding the present study
* Substance abuse
* Inability to follow procedures due to psychological disorders or insufficient knowledge of project language (German)
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Pre-existing regular consumption (>1/week) of erythritol
* Fructose-intolerance
* Pre-existing diet (vegetarian, vegan, gluten-free, lactose-free, caloric restriction, etc.)

EryClot-Pilot:

3 participants

Inclusion criteria:

* Healthy participants 18-55 years upon inclusion
* Normal weight (BMI between 19.0-24.9 kg/m2)
* Informed consent signed by participant

Exclusion criteria:

* Severe acute or chronic diseases
* Pregnancy: although no contraindication, pregnancy might influence metabolic state. Female adolescents who are pregnant or have the intention to become pregnant during the course of the study are excluded. In female participants a urine pregnancy test is carried out upon screening
* Substance abuse, smoking
* Inability to follow procedures due to psychological disorders or insufficient knowledge of project language (German)
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Pre-existing regular consumption (>1/week) of erythritol
* Fructose-intolerance

EryClot:

Inclusion criteria:

* Healthy participants 18-55 years upon inclusion
* Normal weight (BMI between 19.0-24.9 kg/m2)
* Informed consent signed by participant,

Exclusion criteria:

* Severe acute or chronic diseases
* Pregnancy: although no contraindication, pregnancy might influence metabolic state. Female adolescents who are pregnant or have the intention to become pregnant during the course of the study are excluded. In female participants a urine pregnancy test is carried out upon screening
* Substance abuse, smoking
* Inability to follow procedures due to psychological disorders or insufficient knowledge of project language (German)
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Pre-existing regular consumption (>1/week) of erythritol or xylitol
* Pre-existing impairment of blood coagulation/thrombocyte function (e.g., hereditary, regular intake of anti-coagulant agents (e.g., NSAIDs, heparin, warfarin, etc.))

EryClot in vitro

Inclusion criteria:

* Healthy participants 18-55 years upon inclusion
* BMI < 30 kg/m2
* Informed consent signed by participant

Exclusion criteria:

* Severe acute or chronic diseases
* Pregnancy: although no contraindication, pregnancy might influence metabolic state. Female adolescents who are pregnant or have the intention to become pregnant during the course of the study are excluded.
* Substance abuse, smoking
* Inability to follow procedures due to psychological disorders
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Pre-existing regular consumption (>1/week) of erythritol or xylitol
* Pre-existing impairment of blood coagulation/thrombocyte function (e.g., hereditary, regular intake of anti-coagulant agents (e.g., NSAIDs, heparin, warfarin, etc.))

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | Change from baseline to 5 weeks after polyol/sucrose intake
  Insulin resistance as measured by the HOMA Index.
EryClot-Pilot Thrombocyte aggregation | Blood samples at timepoint t= 0, 30, 60, 120, 180 minutes
  Thrombocyte aggregation after consumption of test solution measured with a blood sample
EryClot Thrombocyte aggregation | Blood samples at timepoint t= -60, -1, 30, 60, 120, 180 minutes
  Thrombocyte aggregation after consumption of test solution measured with a blood sample
EryClot in vitro: Platelet responsiveness in human platelet rich plasma | One single fasting blood sample at timepoint t = -10 minutes
  Aggregometry assay after addition of erythritol or xylitol in human platelet rich plasma

SECONDARY OUTCOMES:
Glucose tolerance: Insulin | Change from baseline to 5 weeks after polyol/sucrose intake
  Insulin levels during OGTT
Glucose tolerance: Glucose | Change from baseline to 5 weeks after polyol/sucrose intake
  Glucose levels during OGTT
Glucose tolerance: C-Peptide | Change from baseline to 5 weeks after polyol/sucrose intake
  C-peptide levels during OGTT
Glucose tolerance: Glucagon | Change from baseline to 5 weeks after polyol/sucrose intake
  Glucagon levels during OGTT
Glucose tolerance: Fructosamin | Change from baseline to 5 weeks after polyol/sucrose intake
  Fructosamin levels
Glucose tolerance: HbA1C | Change from baseline to 5 weeks after polyol/sucrose intake
  HbA1C levels
Glucose tolerance: Continuous glucose monitoring average | Change from baseline to 5 weeks after polyol/sucrose intake
  Continuous glucose monitoring for average glucose levels
Glucose tolerance: Continuous glucose monitoring glucose variability | Change from baseline to 5 weeks after polyol/sucrose intake
  Continuous glucose monitoring for glucose variability
Glucose tolerance: Continuous glucose monitoring time within range | Change from baseline to 5 weeks after polyol/sucrose intake
  Continuous glucose monitoring for time within range
Glucose absorption | Change from baseline to 5 weeks after polyol/sucrose intake
  Glucose absorption measured by 3-OMG concetrations during OGTT
Metabolomics | Change from baseline to 5 weeks after polyol/sucrose intake
  Metabolomics in plasma, urine and stool samples, measured by 1H-NMR and Liquid Chromatography-Mass Spectrometry (LC-MS).
Gut microbiota composition | Change from baseline to 5 weeks after polyol/sucrose intake
  The taxonomic and functional profiles of the gut microbiota (stool samples) assessed by metagenomic shotgun sequencing.
Gastrointestinal hormones secretion: GLP-1 | Change from baseline to 5 weeks after polyol/sucrose intake
  Secretion of GLP-1 during OGTT
Gastrointestinal hormones secretion: PYY | Change from baseline to 5 weeks after polyol/sucrose intake
  Secretion of PYY during OGTT
Gastrointestinal hormones secretion: Ghrelin | Change from baseline to 5 weeks after polyol/sucrose intake
  Secretion of Ghrelin during OGTT
Gastrointestinal hormones secretion: CCK | Change from baseline to 5 weeks after polyol/sucrose intake
  Secretion of CCK during OGTT
Food intake | Change from baseline to 5 weeks after polyol/sucrose intake
  Food intake assessed with self-reported food records
Gastrointestinal tolerance | Change from baseline to 3 and 5 weeks after polyol/sucrose intake
  Gastrointestinal tolerance recorded by the "Gastrointestinal Symptoms Rating Scale" (GSRS), 15 items rated on 7 Point Likert-Scale, a higher score means a worse outcome. Maximum score: 90, Minimum score: 0
Body composition: fat mass | Change from baseline to 5 weeks after polyol/sucrose intake
  Body composition assessed by mean of bioimpedance analysis: fat mass in kg
Body composition: fat free mass | Change from baseline to 5 weeks after polyol/sucrose intake
  Body composition assessed by mean of bioimpedance analysis: fat free mass in kg
EryClot-Pilot Blood p-Selectin concentrations | Blood samples at timepoint t= 0, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood p-Selectin concentrations after consumption of test solution
EryClot-Pilot Blood Erythritol concentrations | Blood samples at timepoint t= 0, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood Erythritol concentrations after consumption of test solution
EryClot blood p-selectin concentrations | Blood samples at timepoint t= -60, -1, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood p-Selectin concentrations after consumption of test solution
EryClot blood sVCAM1 concentrations | Blood samples at timepoint t= -60, -1, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood sVCAM1 concentrations after consumption of test solution
EryClot blood PF4 concentrations | Blood samples at timepoint t= -60, -1, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood PF4 concentrations after consumption of test solution
EryClot blood D-Dimers concentrations | Blood samples at timepoint t= -60, -1, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood D-Dimers concentrations after consumption of test solution
EryClot blood Erythritol concentrations | Blood samples at timepoint t= -60, -1, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood erythritol concentrations after consumption of test solution
EryClot blood Xylitol concentrations | Blood samples at timepoint t= -60, -1, 30, 60, 120, 180 minutes and 24, 48 hours
  Blood xylitol concentrations after consumption of test solution

CONTACTS AND LOCATIONS:
Overall Officials: Bettina K. Wölnerhanssen, PD. MD, Principal Investigator — St. Clara Research Ltd.
Locations (1):
- St. Claraspital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No